CLINICAL TRIAL: NCT04474795
Title: Clinic to Community Connections: Enhancing Prenatal to Postpartum Care Transitions to Prevent Type 2 Diabetes in Low Income Women With Gestational Diabetes
Brief Title: Clinic to Community Connections - Broader Distribution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Longer Life Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202007060; 1K23HD096204-01A1 (NIH)
Record Dates: First submitted 2020-05-18; First posted 2020-07-17 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-01

CONDITIONS: Gestational Diabetes; Gestational Diabetes Mellitus in Pregnancy
Keywords: diabetes in pregnancy; type 2 diabetes prevention; diabetes; Care coordination; care delivery; care fragmentation; community health worker; community partnership; community health aides; federally qualified health center; underserved population; patient education
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Staff participants will complete surveys on diabetes knowledge, attitudes, and self-efficacy before and after completing online training modules on gestational diabetes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Staff - Educational training (Experimental): Nurses, community health workers, and others involved in maternal healthcare
  Interventions: Behavioral: Staff -Educational training

INTERVENTIONS:
Behavioral: Staff -Educational training — Nurses and community health workers will complete 4 hours of online modules on gestational diabetes - Module 1: GDM Disease, Diagnosis and Complications; Module 2: Nutrition and Physical Activity Management; Module 3: Monitoring, Medications, and Avoiding Hypoglycemia; Module 4: Future Diabetes Risk and Prevention. Effectiveness of the training will be evaluated with pre/post evaluation of diabetes knowledge, attitudes, and self efficacy.

SUMMARY:
This study addresses education needs in gestational diabetes care and followup at the staff and patient levels.

In the initial phase, nurses and community health workers will complete specific training modules on gestational diabetes developed for this study. The effectiveness of the education modules will be evaluated through pre/post surveys of participants assessing diabetes knowledge, attitudes, and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

Clinic staff: nurses (RN, LPN, BSN), community health workers, and others involved in maternal child health care

Exclusion Criteria:

Clinic staff: individuals not involved in maternal child health care or who do not consent to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J Herrick, MD, MPHS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Affinia Healthcare, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krutilova P, Williams R, Morey R, Field C, Byrth V, Tepe M, McQueen A, Herrick C. Gestational diabetes knowledge improves with interactive online training modules. BMC Med Educ. 2024 Sep 9;24(1):977. doi: 10.1186/s12909-024-05969-z. PMID 39251972
- [Derived] Krutilova P, Williams R, Morey R, Field C, Byrth V, Tepe M, McQueen A, Herrick C. Gestational diabetes knowledge improves with interactive online training modules: a pre-post analysis. Res Sq [Preprint]. 2023 Jun 2:rs.3.rs-2860961. doi: 10.21203/rs.3.rs-2860961/v1. PMID 37398401

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Staff - Educational Training
Started | 85
Completed Pre-test | 82
Accessed Training Module 1 | 65
Accessed Training Module 2 | 45
Accessed Training Module 3 | 41
Accessed Training Module 4 | 20
Completed | 20
Not Completed | 65

BASELINE CHARACTERISTICS:
Population: Population of individuals who completed at least 50% of one of the measures on the baseline survey
Arm/Group | Staff - Educational Training
Number analyzed (Participants) | 82
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37.0 [30.0 to 49.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American, non-Hispanic | 14
  Latinx or Hispanic | 8
  Native American, Asian, another race | 7
  White, non-Hispanic | 53
Region of Enrollment [Number; unit: participants]
  United States | 82
Education/Training [Count of Participants; unit: Participants]
  Nurses (RN/LPN/CHN), CDCES, or RD | 46
  CHW or MA | 18
  Other | 18
Specialty [Count of Participants; unit: Participants]
  Internal Medicine/Family Medicine | 7
  Ob-Gyn/Maternal -Child Health | 52
  Other | 23
GDM knowledge score [Median (Inter-Quartile Range); unit: units on a scale]
  Overall Score | 56.5 [48.4 to 65.2]
  Module 1 Score | 60.0 [60.0 to 80.0]
  Module 2 Score | 66.7 [50.0 to 66.7]
  Module 3 Score | 57.1 [42.9 to 57.1]
  Module 4 Score | 40.0 [40.0 to 60.0]
Self-Efficacy to Provide Diabetes Education Scale [Median (Inter-Quartile Range); unit: units on a scale] | 7.00 [5.90 to 8.27]
Diabetes Attitudes Scale [Median (Inter-Quartile Range); unit: units on a scale]
  Patient autonomy | 4.25 [3.97 to 4.50]
  Value of tight control | 4.14 [3.71 to 4.57]
  Need for special training | 4.80 [4.60 to 5.00]
Intention to Recommend Diabetes Prevention Measures [Median (Inter-Quartile Range); unit: units on a scale] | 4.63 [4.13 to 5.00]

OUTCOME MEASURES:

1. Primary Outcome: Staff - Self-efficacy to Provide Diabetes Education Questionnaire (Newly Developed)
Description: Pre-Post change in staff participants' perceived self-efficacy to provide diabetes education (Mean score min:1 max 10) high score=more confident
Time Frame: Baseline and upon module completion (approximately 3 months)
Population: Population who completed pre and post training assessments and accessed all 4 training modules
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Staff - Educational Training
Number analyzed (Participants) | 20
units on a scale
  Pre-training Score (Baseline) | 6.60 [4.93 to 7.66]
  Post-training Score (Module Completion) | 9.33 [9.00 to 9.87]
Statistical Analysis 1: Comparison: Staff - Educational Training; Compared pre and post training scores; Test type: Superiority; p < 0.0001, Wilcoxon paired signed rank test

2. Secondary Outcome: Staff - Diabetes Knowledge Test
Description: Change in diabetes knowledge measured by multiple choice test (% correct out of 21 items) high score =better knowledge
Time Frame: Baseline and upon module completion (approximately 3 months)
Population: Individuals who completed pre and post-test assessments and accessed all 4 training modules
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Staff - Educational Training
Number analyzed (Participants) | 20
units on a scale
  Pre-training score (Baseline) | 56.5 [48.9 to 65.2]
  Post-training score (Module completion) | 78.3 [65.2 to 87.0]
Statistical Analysis 1: Comparison: Staff - Educational Training; Comparison of scores pre and post training in individuals who completed training modules; Test type: Superiority; p < 0.0001, Wilcoxon paired signed rank test

3. Secondary Outcome: Staff - Diabetes Attitudes (Diabetes Attitudes Scale-3 (DAS-3))
Description: Change in diabetes attitudes measured by 3 subscales of DAS-3 (Mean score min 1, max 5) high score=better attitudes
Time Frame: Baseline and upon module completion (approximately 3 months)
Population: Pre and post training scores in individuals who completed training modules
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Staff - Educational Training
Number analyzed (Participants) | 20
units on a scale
  Pre-training score (Patient Autonomy) | 4.44 [3.75 to 4.59]
  Post-training score (Patient Autonomy) | 4.38 [3.91 to 4.63]
  Pre-training score (value of tight control) | 4.07 [3.75 to 4.54]
  Post-training score (value of tight control) | 4.43 [4.00 to 4.86]
  Pre-training score (need for special training) | 5.00 [4.60 to 5.00]
  Post-training score (need for special training) | 5.00 [4.65 to 5.00]
Statistical Analysis 1: Comparison: Staff - Educational Training; Patient autonomy; Test type: Superiority; p = 0.606, Wilcoxon paired signed rank test
Statistical Analysis 2: Comparison: Staff - Educational Training; Value of tight control; Test type: Superiority; p = 0.003, Wilcoxon paired signed rank test
Statistical Analysis 3: Comparison: Staff - Educational Training; Need for Special Training; Test type: Superiority; p = 0.475, Wilcoxon paired signed rank test

4. Secondary Outcome: Staff - Intention to Recommend Diabetes Prevention Activities Questionnaire (Newly Developed)
Description: Change in staff's intention to recommend postpartum diabetes screening measured by a survey developed for this study (mean score; min 1, max 5) higher score= increased intention to perform action
Time Frame: Baseline and upon module completion (approximately 3 months)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Staff - Educational Training
Number analyzed (Participants) | 20
units on a scale
  Pre-training score | 4.81 [4.37 to 5.00]
  Post-training score | 5.00 [5.00 to 5.00]
Statistical Analysis 1: Comparison: Staff - Educational Training; Test type: Superiority; p = 0.009, Wilcoxon paired signed rank test

5. Other Pre Specified Outcome: Staff-General Self Efficacy Scale (Schwarzer)
Description: General Self Efficacy measure (for use in validation of the Self-Efficacy for Providing Diabetes Education Scale) Sum Score (min: 10, max: 40); higher score=more confidence
Time Frame: Baseline
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Staff-Provider Teaching Motivation Questionnaire Intrinsic Motivation Subscale
Description: Measure of teaching motivation (for use in validation of the Self-Efficacy for Providing Diabetes Education Scale) Mean score (min: 0, max 4) higher score=more intrinsic motivation
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Individuals were not assigned to an intervention that was anticipated to result in adverse events. Individuals had the opportunity to contact the study team with questions or concerns at any time over the course of the study.
Arm/Group | Staff - Educational Training
All-Cause Mortality (participants affected / at risk) | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT04474795/Prot_SAP_000.pdf